CLINICAL TRIAL: NCT00515606
Title: Noninvasive Positive Pressure Ventilation Using Helium:Oxygen Versus Air:Oxygen in Acute Respiratory Failure in Chronic Obstructive Pulmonary Disease Patients Exposed to Sulfur Mustard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 210586
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchiolitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: helium:oxygen

SUMMARY:
to assess the effectiveness of helium:oxygen mixture adjunct with non-invasive ventilation in sulfur mustard exposed patients with acute decompensation

ELIGIBILITY:
Inclusion Criteria:

* a history of previous exposure to sulfur mustard
* worsening dyspnea during the last 10 days
* respiratory rate >25/min
* arterial pH<7.35
* PaCO2 of >50 mmHg
* PaO2 of <50 mmHg

Exclusion Criteria:

* recent pneumothorax (<1 month)
* severe respiratory failure or hemodynamic instability with forthcoming intubation
* FIO2 of <0.4
* impaired consciousness or absence of patient cooperation
* facial lesions precluding NIV

Ages: 38 Years to 59 Years | Sex: Male
Age Groups: Adult
Dates: Start 2007-02; Study Completion 2007-06

PRIMARY OUTCOMES:
assess spirometry and hemodynamic measures after heliox or air:oxygen use

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ghanei, MD, Study Director — Research Center of Chemical Injuries, Baqiyatallah Medical Sciences University